CLINICAL TRIAL: NCT04687423
Title: A Multicenter, Open, Single-arm Phase I Dose Exploration and Phase II Extended Study Was Conducted to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Primary Antitumor Activity of FCN-011 in Patients With Advanced Solid Tumor (Phase I) and NTRK Fusion Positive Advanced Solid Tumor (Phase II)
Brief Title: Study of FCN-011 in Patients With Advanced Solid Tumor（Phase I）and NTRK Fusion Positive Advanced Solid Tumor （Phase II）
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fochon Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-011-001
Record Dates: First submitted 2020-12-10; First posted 2020-12-29 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Advanced Solid Tumor
Keywords: NTRK; FCN-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: phase I dose exploration (Experimental): FCN-011 will be given orally in ascending doses in patients with advanced solid tumor , until the maximum tolerated dose or recommended dose is reached.
  Interventions: Drug: FCN-011

INTERVENTIONS:
Drug: FCN-011 — FCN-011 will be given orally in ascending doses starting at 50 mg Q12h or 100mg QD until the maximum tolerated dose or recommended dose is reached.

SUMMARY:
A multicenter, open, single-arm phase I dose exploration and phase II extended study was conducted to evaluate the safety, tolerability, pharmacokinetic characteristics, and primary antitumor activity of FCN-011 in patients with advanced solid tumor (phase I) and NTRK fusion positive advanced solid tumor (phase II)

DETAILED DESCRIPTION:
This study is a multicenter, open, single-arm Phase I/II clinical study, which is divided into two research parts, namely phase I dose exploration study and phase II dose extension study. In the phase I dose exploration study, the safety, tolerance and PK characteristics of FCN-011 in patients with advanced solid tumors were determined, the MTD of oral fCN-011 was determined, and the RP2D of FCN-011 in the phase II clinical study was determined, and the efficacy of FCN-011 was preliminarily evaluated. The phase II dose extension study evaluated the efficacy, safety, and tolerability of continuous oral ADMINISTRATION of FCN-011 in patients with inoperable NTRK fusion and advanced stage III or IV solid tumors, as well as the characteristics of population pharmacokinetics (PopPK).

A total of 35-82 patients were enrolled in this study, 15-24 patients were expected to be enrolled in the phase I study, and 20-58 patients were expected to be enrolled in the phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years，no gender limitation；
2. Patients with inoperable solid tumors, stage III or IV, confirmed histologically or cytologically by standard treatment failure or no standard treatment;
3. Sufficient tumor tissue samples from clinical phase I patients shall be sent to the central laboratory for NTRK fusion gene test, and the results of the central laboratory will not affect the inclusion of subjects (if multiple patients are screened, patients with positive NTRK fusion gene or point mutation will be preferred to be included);
4. Sufficient tumor tissue samples must be provided for phase II clinical patients, which will be confirmed to be positive for NTRK fusion gene by the method of 2-generation gene sequencing by the central laboratory designated by the sponsor;
5. The ECOG Scores 0 or 1 for physical fitness (phase I),0-2(phase II) ;
6. Can understand and be willing to sign informed consent prior to the commencement of any research procedure; Expected survival at least 12 weeks;
7. Patients with adequate organ and bone marrow function: absolute value of neutrophils ≥ 1.0 × 10^9/L (no G-CSF treatment within 7 days);Hemoglobin ≥ 80g/L (no erythrocyte infusion within 7 days);Platelet ≥ 75 × 10^9/L; Serum total bilirubin ≤ 1.5 × upper limit normal (ULN), and patients with Gilbert syndrome ≤3.0 × ULN. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN; For patients with liver metastasis, AST and ALT should be ≤ 5 × ULN. Creatinine<1.5×ULN or Creatinine clearance was ≥ 60 ml/min in phase I patients, and ≥ 45ml/min in phase II patients. Creatinine clearance was calculated by Cockroft - Gault formula. Albumin ≥ 3g/dL;
8. At least one evaluable lesion (stage I) was assessed according to RECIST 1.1 or RANO criteria; According to RECIST 1.1 or RANO standard to evaluate, at least one measurable lesions (phase II) (primary central nervous system tumors according to the standard definition RANO, needs to have one or more measurable lesions by MRI assessment, size for at least 10 mm or more, and appeared in two or more ≤ 5 mm thick section, the measure does not include cystic cavity.) The imaging evaluation should be completed within 28 days before enrollment, and the patient's hormone dosage should be stable for at least 5 days or more;
9. A fertile woman must have a negative serum pregnancy test within 28 days of the first study drug administration and agree to contraception between 28 days before the first study drug administration and 30 days after the last study drug administration; Male patients are required to undergo ligation or agree to contraception and refuse sperm donation from 7 days before the first dose to 30 days after the last dose; The failure rate of contraceptive methods<1% per year, such as double screen contraceptive methods, condoms, oral or injectable contraceptives.

Exclusion Criteria:

1. Patients who received targeted therapy within 2 weeks or within 5 half-lives (whichever is shorter) before starting administration, and who received chemotherapy, major surgery, radiotherapy, immunotherapy or clinical trials within 4 weeks or within 5 half-lives (which is shorter);
2. Uncontrolled or symptomatic brain metastases (asymptomatic or stably controlled CNS metastases and no hormone therapy within 2 weeks are allowed to be enrolled);Patients with spinal cord metastasis with symptoms of spinal cord compression;Primary CNS tumors were allowed to be enrolled.
3. The toxicity of previous anti-tumor therapy has not recovered (>NCI-CITCAE 5.0 level 2), neurotoxic reaction level 2, except hair loss;
4. Patients should use strong CYP3A4 inhibitors (except drugs permitted in Section 6.8), inducers or sensitive substrates and sensitive substrates of CYP2B6 at the same time;
5. Patients take drugs (mainly Ia, Ic, class III anti-arrhythmia drugs) that will prolong the QTc interval or have risk factors for extending the QTc interval;
6. Difficulty in swallowing, or having an absorbance syndrome, or other medical conditions that prevent the absorption of drugs through the intestinal tract, or affect the absorption of FCN-011;
7. Cardiac function and disease meet one of the following conditions:

（1）screening period in research center 3 times of 12 lead ECG measurement, according to the instrument of QTc formula for calculating the average three times, QTc>470 ms;

（2）continue uncontrolled hypertension, systolic blood pressure under antihypertensive treatment >150 mmHg, and/or diastolic pressure >100 mmHg；

（3）the American New York Heart Association (New York Heart Association, NYHA) classification of grade 3 or more congestive Heart failure;

（4）Arrhythmias of clinical significance, including but not limited to complete left bundle branch conduction anomaly, degree II atrioventricular block;

（5）within 6 months prior to screening of a history of heart attack or a stroke within three months.

8. Phase I with active bacterial, fungal or viral infections of clinical significance, including hepatitis B (hepatitis B virus surface antigen-positive with HBV DNA exceeding 1000 IU/ml) or hepatitis C (HCV RNA positive), human immunodeficiency virus infection (HIV positive);Active bacterial, fungal or viral infections of clinical significance phase II, including patients with chronic hepatitis B with elevated aminotransferase or with evidence of cirrhosis (hepatitis B carriers allowed), positive hepatitis C virus (HCV) antibody test; Confirmed human immunodeficiency virus (HIV) infection and unwillingness to take HIV tests;

9. Has a past or present co-existing malignancies (other than non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignancies that have not been treated and that have been effectively controlled in the past five years) in addition to the indications;

10. Phase II should exclude patients who have previously used TRK gene targeted kinase inhibitor progression, including Entrectinib, Larotrectinib, etc. If the drug is discontinued due to an intolerant toxicity and the duration of treatment is less than 28 days, enrollment is allowed;

11. Patients with known drug-resistant mutations (including but not limited to NTRK1 G595R and NTRK3 G623R) were excluded in phase II;

12. Women who are pregnant or breastfeeding. Any patient who becomes pregnant during the trial should withdraw from the study;

13. Any other disease or condition of clinical significance (such as uncontrolled diabetes, active or uncontrolled infection, etc.) that the investigator considers may affect protocol compliance or affect the patient's signing of the ICF.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
To determine the occurrence of treatment-related adverse events meeting the criteria for dose limiting toxicities (DLTs) | 30 days
The recommended phase II dose for FCN-011 | From first dose up to 30 days after last dose
Overall response rate (ORR) by Response Criteria in Solid Tumors (RECIST) v1.1 | Baseline up to approximately 1 year

SECONDARY OUTCOMES:
To quantify the occurrence of adverse events (AEs) reported in all subjects who received study drug | From enrollment up to 30 days after last dose
the death of the last medicine occurred within 30 days of frequency and cause of death | From enrollment up to 30 days after last dose
The occurrence of treatment-emergent adverse events (TEAs) | From enrollment up to 30 days after last dose
To quantify the last time point with a quantifiable concentration (AUClast) of FCN-011 after administration as a single agen | 2 months
To measure the time to reach the highest plasma concentrations (Tmax) of FCN-011 after single agent administration | 2 months
To quantify the terminal half-life (T1/2) of FCN-011 after administration as a single agent | 2 months
To quantify the dose-dependent serum concentrations (Cmax) of FCN-011 as a single agent | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hu Xi chun, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China